CLINICAL TRIAL: NCT07296796
Title: The Impact of Mindful Compassion on Supporting Women Post-cancer Treatment's Sexual Functioning and Quality of Life in Home Hospice Care: A Preliminary Randomised Controlled Trial.
Brief Title: The Impact of Mindful Compassion on Sexual Functioning and Quality of Life in Home Hospice Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LondonsMU
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sexual Function Disturbances; End of Life; Quality of Life; Well-Being, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Death; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Waitlist controlled study with an active and delayed group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Mindful compassion group provided over 4 weeks
  Interventions: Behavioral: Mindful compassion
- Delayed group (Active Comparator): Mindful compassion group commences at week 4 when the active group intervention terminates.
  Interventions: Behavioral: Mindful compassion

INTERVENTIONS:
Behavioral: Mindful compassion — Participants were encouraged to engage in at home exercises, including breathing exercises, diaries for sexual desire and fantasies, and mindfulness and self-compassion practices such as working on body image. This approach was guided by the 3 system model of emotions, where focusing on the mind and body helps identify physiological changes related to a perceived threat, cognitively recognising and attending to internal and external triggers, and incorporating mindful acceptance and compassion to address the critical inner voice. These techniques will be applied both to daily life and sexual intimacy.

SUMMARY:
Sexual dysfunction is commonly reported post cancer treatments. Indeed, sexual wellbeing can be affected by diagnosis, medication and cancer treatments, which can damage body tissues such as the vagina owing to radiation therapy, or insufficient lubrication caused by chemotherapy. Additionally, feeling sore, exhausted, anxious, depressed and 'not in the mood' further contribute to changes in sexual desire

Very few evidence based online interventions have been developed to address sexual difficulties post cancer treatments and in hospice at home care. This extends to well being and quality of life. Mindful compassion interventions has been based on a behavioural taxonomy to support the reliability of their delivery. Indeed, this study aims to identify and describe the key components and behaviour change techniques as part of the online intervention. These have been mapped to a behaviour change taxonomy with the view of supporting standardisation for future trial implementation. Therefore, the aim of this study is to examine the effectiveness of an online mindful compassion intervention using the 3 system model of emotions among a post cancer treatment group in hospice care, at the end of life, to improve quality of life. The study intends to provide preliminary estimates of pre-post intervention on a waitlist controlled randomised controlled trial looking at well being, sexual function, mindfulness and self compassion.

Quantitatively, the research is structured so that participants will be randomised to either the active experimental or delayed group. This intervention will be weekly for approximately 1 to 2 hours over 4 weeks. This A follow up at 12 weeks will be taken to determine the sustainability of this intervention. Feedback questions will also be given during the delivery of the intervention.

DETAILED DESCRIPTION:
Hospice care is a specialised form of palliative care provided during the later stages of life. Although these two types of care share some similarities, they can differ in timing, location, and available treatments. Hospice care can be delivered at home or in a hospice healthcare centre. While the main treatments are generally discontinued, pain management and support for other health issues, such as high blood pressure or psychological distress like anxiety or depression, may continue. Hospice care, as a component of palliative care, prioritises quality of life and overall well being. Additionally, hospice support can be provided at any point during the patient's condition, not solely in its final stages. A combination of in-home and healthcare support, as well as inpatient care, is also available. Among women, lung cancer, followed by breast cancer, is the most reported cancer in hospice.

The quality of life in palliative care and hospice is vital, given the challenges faced by patients, caregivers, practitioners, families, and partners. It includes overall well being, covering physical, psychological, social, and spiritual aspects. Palliative care provides essential support when addressing the biopsychosocial components of quality of life. However, issues emerge when discussing sex. Despite recognition by organisations such as Marie Curie and Macmillan, there seems to be a reluctance to raise awareness or support research on this topic.

A range of psychosocial interventions is available for individuals after cancer treatment. An increasingly popular approach involves using mindfulness and mindful compassion to support psychosexual functioning. Mindful compassion has been utilised in psychosexual services, including various sexual issues such as sexual pain disorder. Indeed, the three systems model can be used to map out, validate, and normalise different emotional experiences as well as to illustrate how they can influence sexual arousal and enjoyment.

Research on mindfulness and mindful compassion for women after cancer treatments is limited and remains scarce among those in hospice end of life care. This is a sensitive but vital area, as sexual intimacy should not cease with a prognosis. The sense of connection to others is essential at the end of life, and this does not exclude sexual intimacy. This study aimed to assess the effectiveness of an online mindful compassion intervention, based on the 3 system model of emotions, among women with cancer and those receiving hospice care at home.

It was hypothesised that mindful compassion would improve sexual functioning, mindfulness, well-being, and quality of life among women following cancer treatment and in palliative care. Questionnaires were limited because the team did not want to overburden these women, as the focus was on the experience of brief mindful compassion.

ELIGIBILITY:
Inclusion Criteria:

* Were in hospice care with a cancer diagnosis/terminal
* We're receiving support and care
* Identified as female
* Registered with a healthcare service or charity
* Self-perceived satisfactory sexual intimacy before cancer diagnosis (Acquired)
* Aged 18 years or older
* Had a computer, laptop, mobile phone- intervention was online.
* Read and wrote English, as the intervention was delivered in English
* Patient Health Questionnaire 9 screening (score range from minimal to moderate, 0-14).
* Mental Capacity Mini Cog outcomes 3,4,5 (cognitive comprehension)

Exclusion Criteria:

* Were not in hospice care with a cancer diagnosis/terminal
* Did not identify as female
* Were very late-stage palliative/hospice care in which capacity (medication) may be compromised, or discomfort is experienced
* Were aged below 18 years old
* Had reading and writing difficulties in English
* Had a moderate to severe to high Patient Health Questionnaire 9 screening score (ranging from moderate to severe 15-27).
* Mental Capacity Mini Cog outcomes 0,1,2 (problematic cognitive comprehension)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 22 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index | 0, 4 and 12 weeks
  This is a 19 item questionnaire on sexual function, including sexual desire, orgasm, lubrication, sexual satisfaction and pain. It has five response categories. Scores include severe 2-7.2, moderate 7.3-14.4, mild to moderate 14.5-21.6, mild 21.7- 28.1 cut-off value, and no female sexual dysfunction 28.2 -36.The lower the score, the higher the level of sexual dysfunction.
The Short Warwick Edinburgh Mental Wellbeing Scale | 0, 4 and 12 weeks
  A 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of well being. The response categories include 1=none of the time to 5=all of the time. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.
Brief Quality of Life Scale | Weeks 0, 4 and 12
  An 8 item questionnaire with five response categories looking at satisfaction with self, friends, family and creativity. The total score is calculated by summing the satisfaction ratings and summing the six products for a total score with score range between 0-96.
The Self compassion Scale | Weeks 0, 4 and 12
  This is a 12 item measure with five response categories, 1 = almost never to 5= almost always, with higher scores indicating higher levels of self-compassion. The questionnaire measures self-kindness and self-judgement, common humanity and isolation, and mindfulness and over-identification with painful thoughts and emotions. Scores range between. An estimated score between 1-2.5 for overall self-compassion score indicates low levels of self-compassion. 2.5-3.5 indicates moderate. 3.5-5.0 means high levels of overall self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Metropolitan University
Locations (1):
- School of Social Sciences and Professions, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wislawski J, Kasperlik-Zaluska A, Bonicki W, Piotrowska B. [Microadenomas of the pituitary treated by a microsurgical method using the approach through the sphenoid sinus]. Pol Tyg Lek. 1987 Oct 5-12;42(40-41):1266-8. No abstract available. Polish. PMID 3438201
- [Result] Brotto LA, Dunkley CR, Breckon E, Carter J, Brown C, Daniluk J, Miller D. Integrating Quantitative and Qualitative Methods to Evaluate an Online Psychoeducational Program for Sexual Difficulties in Colorectal and Gynecologic Cancer Survivors. J Sex Marital Ther. 2017 Oct 3;43(7):645-662. doi: 10.1080/0092623X.2016.1230805. Epub 2016 Sep 3. PMID 27592509
- [Result] Davison SL. Hypoactive sexual desire disorder. Curr Opin Obstet Gynecol. 2012 Aug;24(4):215-20. doi: 10.1097/GCO.0b013e328355847e. PMID 22729093
- [Result] Jurin T, Sostaric M, Jokic-Begic N, Lauri Korajlija A. mSexHealth: An Overview of Mobile Sexual Health Applications. J Sex Marital Ther. 2023;49(2):129-140. doi: 10.1080/0092623X.2022.2079576. Epub 2022 Jun 2. PMID 35652779
- [Result] Banbury S, Tharmalingam H, Lusher J, Erridge S, Chandler C. A Preliminary Investigation into the Use of Cannabis Suppositories and Online Mindful Compassion for Improving Sexual Function Among Women Following Gynaecological Cancer Treatment. Medicina (Kaunas). 2024 Dec 7;60(12):2020. doi: 10.3390/medicina60122020. PMID 39768900
- [Result] Bagherzadeh R, Sohrabineghad R, Gharibi T, Mehboodi F, Vahedparast H. Effects of mindfulness-based stress reduction training on rumination in patients with breast cancer. BMC Womens Health. 2022 Dec 28;22(1):552. doi: 10.1186/s12905-022-02124-y. PMID 36575482
- [Result] Borson S, Scanlan JM, Chen P, Ganguli M. The Mini-Cog as a screen for dementia: validation in a population-based sample. J Am Geriatr Soc. 2003 Oct;51(10):1451-4. doi: 10.1046/j.1532-5415.2003.51465.x. PMID 14511167
- [Result] Sears C, Millman R, Brotto LA, Walker LM. Feasibility and Acceptability of a Group-Based Mindfulness Intervention for Sexual Interest/Arousal Disorder Following Breast Cancer Treatment. J Sex Marital Ther. 2023;49(5):533-549. doi: 10.1080/0092623X.2022.2154296. Epub 2022 Dec 27. PMID 36573823
- [Result] Smith EJ, Palevsky S. Salt poisoning in a two-year-old child. Am J Emerg Med. 1990 Nov;8(6):571-2. doi: 10.1016/0735-6757(90)90183-z. No abstract available. PMID 2222612
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451